CLINICAL TRIAL: NCT02343783
Title: A Phase 0 Study Exploring the Use of Induced Skin Blisters in Adult Subjects With Atopic Dermatitis, Allergic Asthma and Atopic Healthy Subjects.
Brief Title: A Study to Evaluate Use of Induced Skin Blisters in Adult Participants With Atopic Dermatitis, Allergic Asthma and Atopic Healthy Participants
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR106398; NOCOMPOUNDNAP0005 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-01-16; First posted 2015-01-22 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Dermatitis, Atopic; Asthma; Healthy
Keywords: Atopic Dermatitis; Asthma; Healthy; Skin Blisters; Adult Participants
MeSH Terms: conditions — Dermatitis, Atopic; Asthma; Blister

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy + Atopic Dermatitis + Allergic Asthmatic Participants (Experimental): Healthy participants will be enrolled in order to allow for training on the overall skin blister induction and fluid aspiration process. Participants with atopic dermatitis (AD) or allergic asthma (AA) will be observed for the use of induced skin blisters after allergic skin reaction (ASR).
  Interventions: Other: Allergic Skin Reaction (ASR) Testing and Skin Blister Induction

INTERVENTIONS:
Other: Allergic Skin Reaction (ASR) Testing and Skin Blister Induction — Participants will not receive any intervention in this study. Healthy participants will be enrolled in order to allow for training on the overall skin blister induction and fluid aspiration process. The cell populations and inflammatory mediator responses in suction skin blister fluid after allergic skin reaction (ASR) in participants with atopic dermatitis (AD) or allergic asthma (AA) will be observed.

SUMMARY:
The purpose of this study is to characterize the cell (the basic building block of all living things) populations and inflammatory (pain and swelling) mediator responses in suction skin blister fluid after allergic skin reaction (ASR) [rash] induction with D. Pteronyssinus [house dust mite (HDM)], Alternaria alternata, or Aspergillus fumigatus allergens in participants with atopic dermatitis (AD) [Skin rash, Eczema] or allergic asthma (AA) [breathing disorder in which there is a wheezing and difficulty breathing].

DETAILED DESCRIPTION:
This is an interventional (a treatment given during the course of a research study) and multicenter (when more than one hospital or medical school team work on a medical research study) study. The study will consist of 3 Phases: Screening Phase (Up to 4 weeks), Data Collection Phase (9 days) and, Follow-up Phase (7 days). The maximum study duration for each participant will not exceed 43 days. Primarily, the cell populations and inflammatory mediator responses in suction skin blister fluid after allergic skin reaction (ASR) will be assessed. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have signed an informed consent document prior to any study related procedures indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study
* Participant must be willing/able to adhere to the study visit schedule and other requirements, prohibitions and restrictions specified in this protocol

  * For participants with Asthma:
* Participant must have a physician documented diagnosis of asthma for at least 12 months before Screening
* Participant must have an Asthma Control Questionnaire 6 (ACQ6) less than (<) 1.5 at Screening

  * For participants with Atopic Dermatitis:
* Participant must have a physician documented diagnosis of atopic dermatitis for at least 12 months before Screening based on UK refinement of the Hanifin and Rajka's diagnostic criteria
* Participant must have atopic dermatitis with and Investigators Global Assessment (IGA) score of 2 to 4 at Screening

Exclusion Criteria:

* Participant has taken any prohibited or restricted medications as noted below under Prestudy and Concomitant Therapy
* Participant has received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 6 weeks or 5 half-lives (whichever is longer) before the Screening visit

  * For participants with Asthma:
* Participant has a history of life-threatening asthma, defined as a history of respiratory arrest or requiring intubation for asthma
* Participant had been admitted to a hospital for asthma in the 1 year before Screening

  * For participants with Atopic Dermatitis:
* Participant has evidence of any other skin condition that would interfere with assessment of Atopic Dermatitis (AD)
* Participant has active AD related infection or has had an active AD infection within 2 weeks of Screening (participants with evidence of colonization on skin swab testing but with no infection are allowed)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Cell Concentration in Suction Skin Blister Fluid After Allergic Skin Reaction (ASR) Induction with D. Pteronyssinus (House Dust Mite [HDM]), Alternaria alternata, or Aspergillus fumigatus Allergens | Hour 4 after the end of the blister induction
  Cells in the aspirated skin blister fluid will be separated and processed for cell population analysis by flow cytometry and messenger RNA (mRNA) analysis.
Cell Concentration in Suction Skin Blister Fluid After ASR Induction with D. Pteronyssinus (House Dust Mite), Alternaria alternata, or Aspergillus fumigatus Allergens | Hour 24 after the end of the blister induction
  Cells in the aspirated skin blister fluid will be separated and processed for cell population analysis by flow cytometry and mRNA analysis.
Levels of Inflammatory Mediators in Suction Skin Blister Fluid After ASR Induction with D. Pteronyssinus (House Dust Mite), Alternaria alternata, or Aspergillus fumigatus Allergens | Hour 4 after the end of the blister induction
  The remaining fluid from aspirated skin blister fluid after separated and processed for cell population analysis will be assessed for inflammatory mediator responses. Inflammatory cytokines and other soluble mediators in blister fluid will be measured by immunoassay.
Levels of Inflammatory Mediators in Suction Skin Blister Fluid After ASR Induction with D. Pteronyssinus (House Dust Mite), Alternaria alternata, or Aspergillus fumigatus Allergens | Hour 24 after the end of the blister induction
  The remaining fluid from aspirated skin blister fluid after separated and processed for cell population analysis will be assessed for inflammatory mediator responses. Inflammatory cytokines and other soluble mediators in blister fluid will be measured by immunoassay.

SECONDARY OUTCOMES:
Success Percentage of Repeated Skin Blister Induction and Blister Fluid Aspiration | Day 1 and 8
  Success percentage for blister induction will be defined as number of blisters formed with recovery of at least 200 microliter (μL) of blister fluid, divided by the total blisters induced.
Cell Concentration in Suction Skin Blister Fluid After ASR Induction with Non-protease Allergens | 4 and 24 Hours after the end of the blister induction
  Cells in the aspirated skin blister fluid will be separated and processed for cell population analysis by flow cytometry and mRNA analysis.
Levels of Inflammatory Mediators in Suction Skin Blister Fluid After ASR Induction with Non-protease Allergens | 4 and 24 Hours after the end of the blister induction
  The remaining fluid from aspirated skin blister fluid after separated and processed for cell population analysis will be assessed for inflammatory mediator responses. Inflammatory cytokines and other soluble mediators in blister fluid will be measured by immunoassay.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (7):
- Belgium (2):
  - Antwerp
  - Merksem
- Germany (5):
  - Berlin
  - Hamburg
  - Hanover
  - Kiel
  - Mönchengladbach